CLINICAL TRIAL: NCT02649231
Title: A Phase II, Randomised, Double-blind, Placebo- Controlled, Multi-site, Parallel Group Clinical Trial to Examine Ketamine as a Pharmacological Treatment for Alcohol Dependence in an Alcohol Dependent Population
Brief Title: Ketamine for Reduction of Alcoholic Relapse
Acronym: KARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13/0253.
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Results first posted 2021-09-09 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Primary Alcohol Use Disorder
MeSH Terms: interventions — Ketamine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ketamine+Psychological Therapy (Experimental): Ketamine with psychological therapy
  Interventions: Drug: Ketamine; Behavioral: Psychological Therapy
- Ketamine+Education (Active Comparator): ketamine with alcohol education
  Interventions: Drug: Ketamine; Behavioral: Alcohol Education
- Placebo+Psychological Therapy (Active Comparator): placebo with psychological therapy
  Interventions: Drug: Placebo; Behavioral: Psychological Therapy
- Placebo+Education (Placebo Comparator): placebo with simple alcohol education
  Interventions: Drug: Placebo; Behavioral: Alcohol Education

INTERVENTIONS:
Drug: Ketamine — 0.8 mg/kg ketamine
  Arms: Ketamine+Education; Ketamine+Psychological Therapy
Drug: Placebo — 0.9% saline
  Arms: Placebo+Education; Placebo+Psychological Therapy
Behavioral: Psychological Therapy — Manualised relapse prevention based CBT
  Arms: Ketamine+Psychological Therapy; Placebo+Psychological Therapy
Behavioral: Alcohol Education — Simple education about alcohol effects
  Arms: Ketamine+Education; Placebo+Education

SUMMARY:
96 recently detoxified alcoholics will be randomized to receive either 3 sessions ketamine (0.8 mg/kg IV over 45 minutes) or placebo plus manualised psychological therapy, or 3 sessions of ketamine or placebo plus simple psychoeducation. Patients will be assessed at 3 and 6 months on a range of psychological and biological variables. Primary endpoints will be % days abstinent at 6 months and relapse rates at 6 months. Secondary endpoints include depressive symptoms, craving, quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Meet either a) DSM-5 criteria for severe alcohol use disorder and b) DSM-IV criteria for alcohol dependence within the last 12 months;
* Currently abstinent from alcohol (breathalyser BAC level 0.00) and negative urine drug screening (participants testing positive for THC who do not have a history or current cannabis dependency may be included);
* Minimum of mild depression(>14 on Beck Depression Inventory-II);
* Capacity to give informed consent as defined by GCP guidelines;
* Willing and able to wear SCRAM-X bracelet for 6 months;
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; True abstinence) from the time consent is signed until 6 weeks after treatment discontinuation and inform the trial if pregnancy occurs. For the purpose of clarity, True abstinence is when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence, withdrawal, spermicides only or lactational amenorrhoea method for the duration of a trial, are not acceptable methods of contraception;
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for trial treatment and on day of first treatment.

Exclusion Criteria:

* Currently taking any other relapse prevention medication or anti-depressants;
* Uncontrolled hypertension, systolic 140mm Hg or greater and diastolic 90mm Hg or greater;
* <16 or > 35 BMI
* History of psychosis, or in a first-degree relative as identified by DSM-5 or DSM-IV SCID; co-morbid current psychiatric diagnosis excluding depression, identified via self-reported or identified by a medical professional;
* Previous or current diagnosis of substance dependence / severe substance misuse disorder;
* History of neuropsychological difficulties
* One or more previous confirmed seizures;
* Currently taking daily prescribed medication contraindicated in the SPC with ketamine:

  1. Barbiturates and/or narcotics
  2. Atracurium and tubocurarine
  3. Central nervous system (CNS) depressants (e.g. phenothiazines, sedating H1 - blockers or skeletal muscle relaxants)
  4. Anxiolytics, sedatives and hypnotics
  5. Thiopental, thyroid hormones
  6. Antihypertensive agents
  7. Theophylline and methylxanthines.
  8. Halogenated anaesthetics
  9. OR psychotropic drug use at screening assessments or during treatment weeks
* Liver function tests > 3 times normal levels
* Where there are "special warnings or precautions for use" according to the SPC and where risk vs benefit ratio is not in favour of giving ketamine, with assessment made by physical examination by medically qualified trial personnel, self-report or inspection of the medical notes:

  1. Acute intermittent porphyria
  2. Dehydration or hypovolemia
  3. Hyperthyroidism, or patients receiving thyroid replacement
  4. Pulmonary or upper respiratory tract infection
  5. Severe Coronary artery disease, Cerebrovascular accident or cerebral trauma
  6. Diabetes
  7. Known glaucoma or globe injuries
  8. Cirrhosis
  9. Epilepsy
  10. Neurological condition/brain damage
  11. Intracranial mass lesions, presence of head injury or hydrocephalus
* Suicidal ideation.
* Not willing to use effective contraception or (females) take pregnancy test;
* Allergic reaction to ketamine;
* >10 previous detoxifications from alcohol;
* Pregnant or breastfeeding;
* Allergies to excipients of IMP or placebo;
* Use of another experimental investigational medicinal product that is likely to interfere with the study medication within 3 months of study enrolment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celia Morgan, Ph.D., Principal Investigator — UCL
Locations (2):
- United Kingdom (2):
  - NIHR Exeter Clinical Research Facility, Exeter
  - NIHR UCLH Clinical Research Facility, London

REFERENCES:
- [Derived] Grabski M, McAndrew A, Lawn W, Marsh B, Raymen L, Stevens T, Hardy L, Warren F, Bloomfield M, Borissova A, Maschauer E, Broomby R, Price R, Coathup R, Gilhooly D, Palmer E, Gordon-Williams R, Hill R, Harris J, Mollaahmetoglu OM, Curran HV, Brandner B, Lingford-Hughes A, Morgan CJA. Adjunctive Ketamine With Relapse Prevention-Based Psychological Therapy in the Treatment of Alcohol Use Disorder. Am J Psychiatry. 2022 Feb;179(2):152-162. doi: 10.1176/appi.ajp.2021.21030277. Epub 2022 Jan 11. PMID 35012326
- [Derived] Grabski M, Borissova A, Marsh B, Morgan CJA, Curran HV. Ketamine as a mental health treatment: Are acute psychoactive effects associated with outcomes? A systematic review. Behav Brain Res. 2020 Aug 17;392:112629. doi: 10.1016/j.bbr.2020.112629. Epub 2020 May 30. PMID 32485203
- [Derived] McAndrew A, Lawn W, Stevens T, Porffy L, Brandner B, Morgan CJ. A proof-of-concept investigation into ketamine as a pharmacological treatment for alcohol dependence: study protocol for a randomised controlled trial. Trials. 2017 Apr 4;18(1):159. doi: 10.1186/s13063-017-1895-6. PMID 28372596

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo+Education: placebo with alcohol education
  Placebo: 0.9% saline
  Alcohol Education: Simple education about alcohol effects
Period: Overall Study
Arm/Group | Ketamine+Psychological Therapy | Ketamine+Education | Placebo+Psychological Therapy | Placebo+Education
Started | 24 | 24 | 23 | 25
Completed | 20 | 21 | 21 | 23
Not Completed | 4 | 3 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine+Psychological Therapy | Ketamine+Education | Placebo+Psychological Therapy | Placebo+Education | Total
Number analyzed (Participants) | 24 | 24 | 23 | 25 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (8.7) | 40.5 (11.1) | 47.0 (11.8) | 43.7 (10.2) | 44.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 8 | 10 | 35
  Male | 14 | 17 | 15 | 15 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24 | 24 | 23 | 25 | 96

OUTCOME MEASURES:

1. Primary Outcome: Relapse Rates
Description: Time line follow back
Time Frame: 6 months
Population: To explain discrepancies between overall number of participants analysed and the flow diagram: Only participants with a minimum of 159 days of completed drinking self-report data were included in the main analysis of alcohol relapse status as this was the shortest duration of time before any participant completed the 6 month (23-25 week) follow up in the study. Reporting time was capped at 180 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine+Psychological Therapy | Ketamine+Education | Placebo+Psychological Therapy | Placebo+Education
Number analyzed (Participants) | 21 | 22 | 21 | 23
Participants | 13 | 15 | 14 | 18
Statistical Analysis 1: Comparison: Ketamine+Psychological Therapy vs Ketamine+Education vs Placebo+Psychological Therapy vs Placebo+Education; Confirmed alcohol relapse by drug condition at 6 months using the Alcohol Timeline-Followback. Logistic regression modelling was used to compare the ketamine group with the placebo group (combined across therapy and alcohol education); Test type: Superiority; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.28 to 1.75]

2. Primary Outcome: Percentage Days Abstinent
Description: Time line follow back
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Ketamine+Psychological Therapy | Ketamine+Education | Placebo+Psychological Therapy | Placebo+Education
Number analyzed (Participants) | 24 | 24 | 23 | 25
percentage of days abstinent | 86.4 (17.7) | 82.5 (20.0) | 78.3 (26.9) | 70.7 (25.1)
Statistical Analysis 1: Comparison: Ketamine+Psychological Therapy vs Ketamine+Education vs Placebo+Psychological Therapy vs Placebo+Education; Linear regression modelling was used to compare the ketamine group with the placebo group (combined across therapy and psychoeducation). Only participants with a minimum of 159 days of completed drinking self-report data were included in the main ITT analysis as this was the shortest duration of time before any participant completed the 6 month (23-25 week) follow up in the study. Reporting time was capped at 180 days; Test type: Superiority; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [1.1 to 19.0]

ADVERSE EVENTS:
Time Frame: Screening visit (visit 1) to 6 month follow-up visit (visit 10).Participants were asked about any potential adverse events at the beginning of each visit.
Description: Participants were asked about any potential adverse events at the beginning of each visit.
Arm/Group | Ketamine+Psychological Therapy | Ketamine+Education | Placebo+Psychological Therapy | Placebo+Education
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 2/23 | 1/25
Other Adverse Events (participants affected / at risk) | 13/24 | 17/24 | 16/23 | 17/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine+Psychological Therapy (N=24) | Ketamine+Education (N=24) | Placebo+Psychological Therapy (N=23) | Placebo+Education (N=25)
Brain hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Abdominal pain secondary to spontaneous abortion
Alcohol intoxication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine+Psychological Therapy (N=24) | Ketamine+Education (N=24) | Placebo+Psychological Therapy (N=23) | Placebo+Education (N=25)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Arm pain (Surgical and medical procedures) | 1 (2) | 1 (1) | 0 (0) | 0 (0) — Pain in arm were cannula was administered/ blood was taken from.
Dental implantation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction insect bites (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 6 (10) | 0 (0) | 4 (7)
Influenza (General disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Insomnia (General disorders) | 2 (4) | 2 (4) | 2 (2) | 2 (4)
Mental confusion (General disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
Unsteadiness (General disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Lack of coordination (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ankle pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Elbow pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Knee pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Stomach pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toe pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cannula (for infusion) blocked (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 1 (1) | 3 (3) | 3 (3)
Depressed mood (Psychiatric disorders) | 4 (5) | 12 (15) | 7 (8) | 6 (7)
Anger (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Emotional distress during talking session (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Emotionally unstable (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feelings of altered reality (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flat affect (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Loss of interest in activities (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood fluctuations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Passive suicidal thoughts (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure during alcohol withdrawal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tearfulness (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Erection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — During infusion
Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
Anaesthetic shivers (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Broken thumb (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cut heel (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Caused by SCRAM device
Cut finger (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cut at wrist (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Accident
Scratch to forehead (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — After fall
Finger fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hospitalisation due to morphine overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
IV cannula infiltration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sprained ankle (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Whiplash associated disorder (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Viral rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 2 (3) | 4 (4)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coughing up blood (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALT and AST increase in blood test (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia diagnosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Low folic acid (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen glands (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (6) | 4 (5) | 2 (2) | 8 (15)
Impaired concentration (Nervous system disorders) | 0 (0) | 4 (6) | 1 (1) | 2 (3)
Memory impairment (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Altered Time perception (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bodily numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration to forehead due to fall during seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vasovagal syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual distortions (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thirst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin rash arm (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Skin rash leg (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Two red bumps around eyes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain thorax (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strained gluteus maximus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stiff neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Herpes labialis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Finger infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Both hands
Mouth ulcer (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT02649231/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT02649231/SAP_001.pdf